CLINICAL TRIAL: NCT04290026
Title: Ultrasound Assessment of the Effect of Metoclopramide Versus Granisetron on Gastric Volume in Patients Undergoing Caesarean Section
Brief Title: Granisetron Versus Metoclopramide Effects on Gastric Volume by Sonographic Assessment on Patients Undergoing Caesarean Section.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed, Assistent lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: us, gastric volume
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Aspiration Vomitus
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metoclopramide versus granisetron (Active Comparator): Ultrasound assessment of the effect of metoclopramide versus granisetron on gastric volume in patients undergoing caesarean section: A randomized, double-blind, placebo-controlled study
  Interventions: Drug: metoclopramide versus granisetron

INTERVENTIONS:
Drug: metoclopramide versus granisetron — ِِِِAssessment of the effect of metoclopramide versus granisetron on gastric volume in patients undergoing caesarean section by us

SUMMARY:
Ultrasound assessment of the effect of metoclopramide versus granisetron on gastric volume in patients undergoing caesarean section study

DETAILED DESCRIPTION:
Nausea and vomiting in the perioperative period are common sequelae during abdominal operations, with variable rates up to 80%, as reported in the literature. Perioperative nausea and vomiting associated with pregnancy originate from multiple factors. Pregnancy hormones induced lowering of the lower oesophageal sphincter tone, elevated gastric pressure by the effect of gravid uterus, hypotension, manipulation of the uterus during the operation that leads to visceral stimulation, and the use of opioids; which represent some of the proposed causative factors .

There is a lack of cost-effectiveness and consensus about prophylactic antiemetic use before abdominal surgeries. However, there is enough data reported in the literature that suggests the prophylactic use of antiemetic therapy for patients undergoing cesarean section (CS) under either general or regional anesthesia and as rescue medication for the treatment of episodes of intraoperative and postoperative nausea and vomiting.

Metoclopramide studied intensively as one of the best premedications in patients undergoing abdominal surgeries, especially in the obstetric population. It has a favorable effect on reducing the gastric fluid volume during the operation and consequently decreasing the incidence of aspiration pneumonia .

Granisetron is a selective 5-HT3 receptor antagonist with little or no affinity for other serotonin receptors is classified as drug group B in pregnant patients and approved by the FDA (Food and Drug Administration) for the treatment of post-operative nausea and vomiting in adults . 5-HT3 receptor antagonists exert appropriate clinical efficacy and low incidence of adverse drug reactions. In comparison with ondansetron, granisetron is a more potent antagonist with a longer duration of action .

Different methods such as paracetamol absorption, polyethylene glycol dilution (PEG), and electric impedance tomography (EIT) suggested as methods for visualizing the structure, volume, and time to the emptying of the stomach. Gastric scintigraphy remains the gold standard for such detections . However, scintigraphy is discouraged in routine clinical settings and pregnant patients owing to the risk of radiation exposure, low cost-effectiveness, and intricate instrumental setups.

Gastric ultrasonography (GUS) has emerged as an accessible, cost-effective, safe, and portable diagnostic modality for visualizing the gastric morphology. Different studies suggest that gastric contents and volume measured through GUS significantly correlated to the cross-sectional antral area. As a result, the reliability and reproducibility of bedside GUS cannot be challenged.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age :18-45
* Informed consent

Exclusion Criteria:

1. women who have a history of :

   * diabetes mellitus
   * hypertension
   * preeclampsia
   * neurological and psychological disorders
   * renal or hepatic diseases
   * chronic Gerd
2. refusal to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — patients undergoing caesarean section
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
1. The size of the cross-sectional antral area | Immediately after the procedure
  G-0: Antrum was flat and empty in a supine and right lateral position G-1: Antrum had fluid in the right lateral position but empty in the supine position G-2: Antrum had fluid and food in both the supine and right lateral position.

SECONDARY OUTCOMES:
The incidence of post operative nausea or vomiting and the effects on the hemodynamic status | 1day

CONTACTS AND LOCATIONS:
Overall Officials: saeid metwally, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: 3 years
Access Criteria: age, sex ,clinical diagnosis